CLINICAL TRIAL: NCT06333392
Title: Total Underwater Colonoscopy (TUC) for Improved Colorectal Cancer Screening: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Ullevaal University Hospital (Other); Sahlgrenska University Hospital (Other); Ostfold Hospital Trust (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TotalUnderwater_REK577567
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Neoplasia; Screening Colonoscopy; Colorectal Cancer; Colorectal Cancer Screening; Vasovagal Reaction
Keywords: colorectal cancer screening; screening colonoscopy; underwater colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional colonoscopy (CO2) group (Active Comparator): this groups receives conventional colonoscopy with CO2 withdrawal
  Interventions: Procedure: Conventional colonoscopy
- Total underwater colonoscopy (TUC) group (Experimental): This group receives total underwater colonoscopy
  Interventions: Procedure: Total underwater colonoscopy

INTERVENTIONS:
Procedure: Total underwater colonoscopy — one grooup will be randomized to receive a total underwater colonoscopy
  Arms: Total underwater colonoscopy (TUC) group
Procedure: Conventional colonoscopy — one group will be randomized to undergo a conventional colonoscopy with CO2 withdrawal
  Arms: Conventional colonoscopy (CO2) group

SUMMARY:
Colorectal cancer (CRC), the third most diagnosed cancer and second most common cause of cancer death. CRCs develop from precursors like adenomas (about 70% of CRCs) or serrated lesions (SSLs) (about 25-30% of CRCs). Colonoscopy is the cornerstone in CRC screening, in screening programmes often as a work-up examination after a positive primary screening test such as faecal immunochemical test (FIT). Norway and Sweden have recently launched a nationwide faecal haemoglobin CRC screening programmes. Recently, both a Dutch and an Austrian study showed that SSL detection rate (SSLDR) is inversely correlated to CRC at follow-up. Consequently, improved SSLDR can reduce the risk of post-colonoscopy CRC. SSLs are typically located in the right colon. They are flat, with indistinctive boarders, and consequently easily missed or incompletely resected. A Norwegian study showed incomplete resection of 40% of proximal SSLs. The prevalence of SSLs is higher in women than in men, with women being on a threefold risk of developing CRC from SSLs. It seems like post-colonoscopy CRC more often is caused by SSLs than by adenomas. Total underwater colonoscopy (TUC) is a technique replacing conventional CO2 insufflation by water infusion to distend the lumen and visualise the mucosa during withdrawal of the colonoscope and simultaneously removal of water. There are several reasons to advocate TUC:

1. SSLs will be more visible as they "float" on the submucosa and contract into the lumen, while full distension by gas stretches the mucosa, making detection of flat lesions more difficult.
2. Water works like a magnifying lens, making detection and detailed characterisation of lesions easier.
3. uEMR is eased.
4. Improved bowel cleansing

The goal of this clinical trial is to compare colonoscopy outcomes for standard gas (CO2) insufflation and TUC during withdrawal in patients participating in colonoscopy in the Norwegian and Swedish colorectal cancer screening programme after a positive fecal immunochemical test.

The overarching research questions of the present trial is whether colonoscopy outcomes are improved when CO2 insufflation is replaced by TUC during withdrawal and whether the new technique reduces the ecological footprint of the colonoscopy examination.

The project has five main hypotheses:

1. TUC is superior to the standard approach (CO2 withdrawal) regarding detection of proximal SSLs.
2. TUC increases the rate of complete resection of lesions >= 10mm.
3. TUC reduces the rate of painful colonoscopies and vasovagal reactions.
4. TUC reduces the health care costs by reduced use of single use accessories and reduced number of redundant colonoscopies to obtain polypfree colon.
5. TUC reduces the carbon footprint by reduced use of single use accessories.

If TUC is superior to gas insufflation, the technique may be implemented rapidly since the technique is easy to learn. This study will increase endoscopy competence at participating centres. The centres are involved in national colonoscopy training programs, so the technique will quickly be passed on to other hospitals and screening centres.

The trial can be linked to three of the Global Goals:

* Good health and well-being: The increased detection and improved complete removal of sessile serrated lesions can subsequently decrease the risk of CRC and CRC mortality during follow-up. TUC will probably reduce the rate of painful procedures and vasovagal reactions and thus increase the acceptance of a screening programme. Consequently, the project can contribute significantly to improve screening effectiveness in Norway and Sweden, particularly in women (women have a higher risk for SSLs and a higher risk of colorectal cancer developing from this type of precursor).
* Gender equality: Women have a similar lifetime risk for CRC as men but less benefit of screening regardless of whether they are screened by sigmoidoscopy, FIT or colonoscopy. The reason is probably missed sessile serrated lesions in the proximal colon. If TUC improves SSLDR and complete lesion resection, this may lead to an equal benefit from CRC screening for women and men. Women have also a higher risk of discomfort and pain during colonoscopy than men. It has been shown that women prefer non-invasive screening modalities, potentially to avoid pain during colonoscopy, even if colonoscopy may be the most beneficial screening method for women. If TUC reduces the rate of painful colonoscopies, it can reduce women's barriers to attend screening.
* Responsible consumption and production: The TUC technique will also reduce the ecological footprint of colonoscopy activity due to reduced consumption of single use accessories and reduced number of colonoscopies to achieve polyp free colon. Furthermore, the cost for the health care system will be substantially reduced.

ELIGIBILITY:
Inclusion Criteria:

* All individuals referred to colonoscopy after a positive FIT screening at the participating screening centres

Exclusion Criteria:

* Individuals with a CRC diagnosis within the last 10 years.

Ages: 55 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1070 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proximal sessile serrated lesion detection rate | when histopathology report is clear, about 4 weeks after colonoscopy
  The proportion of colonoscopies where at least one proximal SSL is detected

SECONDARY OUTCOMES:
Complete resection rate for lesions > 10mm | 4 weeks after colonoscopy
  see above
Rate of painful procedures and vasovagal reactions | during and immediately after colonoscopy
  se above
Leakage after colonoscopy | Questionnaire 1-7 days after colonoscopy
  water leakage on the way home after colonoscopy
Detection rate for other neoplasia than SSL | about 4 weeks after colonoscopy
  see above
Withdrawal time | immediately after colonoscopy
  see above
Total procedure time | immediately after colonoscopy
  see above
Bowel cleansing quality | immediately after colonoscopy
  with help of BBPS
Complications | within 30 days after colonoscopy
  Significant bleedings and perforations
Number of colonoscopies to achieve polyp free colon | after last colonoscopy per patient
  see above
Single use accessories for the procedure | immediately after colonoscopy
  number of single use accesoires per colonoscopy
Willingness to repeat colonoscopy | questionnaire 1-2 weeks after colonoscopy
  Willingness to repeat colonoscopy the same way if new colonoscopy is necessary

CONTACTS AND LOCATIONS:
Locations (5):
- Norway (4):
  - Vestre Viken Health Trust, Bærum Hospital, Drammen
  - Østfold Hospital Health Trust, Grålum
  - Akershus University Hospital Health Trust, Lørenskog
  - Ullevål University Hospital Health Trust, Oslo
- Sahlgrenska University Hospital, Gothenburg, Region Västra Götaland, Sweden, Department of Medicine, Geriatrics and Emergency Care Mölndal, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: Access to research data for external investigators, or use outside of the current protocol, will require approval from the Norwegian Regional Committee for Medical and Health Research Ethic. Research data are not openly available because of the principles and conditions set out in articles 6[1] (e) and 9 [2] (j) of the General Data Protection Regulation (GDPR).
URL: http://notavailableyet.no